CLINICAL TRIAL: NCT02004340
Title: Transcutaneous Auricular Vagus Nerve Stimulation as a Complementary Treatment for Pediatric Epilepsy
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation for Pediatric Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Beijing Tiantan Hospital (Other); Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Wei He, Associate Professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSFC-81273829; 2011CB505201 (Other Grant/Funding Number: National Basic Resaearch Program (973 Program))
Record Dates: First submitted 2013-11-13; First posted 2013-12-09 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Epilepsy
Keywords: pediatric epilepsy; transcutaneous vagus nerve stimulation
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Transcutaneous auricular vagal stimulation (Active Comparator): Transcutaneous stimulation at auricular concha
  Interventions: Device: ear vagus nerve stimulator
- Transcutaneous auricular non-vagal stimulation (Sham Comparator): Transcutaneous stimulation at auricular edge
  Interventions: Device: ear vagus nerve stimulator
- control (No Intervention): No transcutaneous stimulation is given

INTERVENTIONS:
Device: ear vagus nerve stimulator
  Arms: Transcutaneous auricular non-vagal stimulation; Transcutaneous auricular vagal stimulation

SUMMARY:
The purpose of this study is to determine whether transcutaneous auricular vagus nerve stimulation as a complementary therapy is effective in the treatment of pediatric epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as epilepsy;
* With age between 2-18 years old;
* The number and dose of the medication was kept constant no less than eight weeks before intervention;
* The patients or their guardians can count the frequency of the seizures and finish the study.

Exclusion Criteria:

* The patient is receiving the VNS therapy;
* Accompanied with progressive central nervous system diseases;
* Have severe heart, liver ,kidney or blood diseases;
* Be pregnant or having the schedule of pregnancy in the study period.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
frequency of epileptic seizures | Change from baseline at 8, 16, 24 weeks respectively in frequency of epileptic seizures

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | participants will be followed for the duration of TVNS intervention, an expected average of 8 weeks"

CONTACTS AND LOCATIONS:
Overall Officials: Bing Zhu, Dr., Study Director — Institute of Acupuncture and Moxibustion, CACMS
Locations (1):
- Wei He, Beijing, China

REFERENCES:
- [Derived] He W, Wang XY, Zhou L, Li ZM, Jing XH, Lv ZL, Zhao YF, Shi H, Hu L, Su YS, Zhu B. Transcutaneous auricular vagus nerve stimulation for pediatric epilepsy: study protocol for a randomized controlled trial. Trials. 2015 Aug 21;16:371. doi: 10.1186/s13063-015-0906-8. PMID 26292720